CLINICAL TRIAL: NCT01388738
Title: Navigation Brain Stimulation (NBS) for Evaluation of the Neuroprotective Drug Efficiency in Patients After Ischemic Stroke.
Brief Title: Navigation Brain Stimulation for Evaluation of the Neuroprotective Drug Efficiency in Patients After Ischemic Stroke.
Acronym: 3C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinical Institute of the Brain, Russia (Other)
Collaborators: Nycomed (Industry); Veropharm (Industry); Ever Neuro Pharma GmbH (Industry)
Responsible Party: prof. Andrey A. Belkin, MD, PhD, Clinical Institute of the Brain, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CIB-NBS-C
Record Dates: First submitted 2011-06-27; First posted 2011-07-07 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Stroke
Keywords: Navigation Brain Stimulation (NEXSTIM); cerebroprotective drug effectiveness; acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Cytidine Diphosphate Choline; Glycerylphosphorylcholine; cerebrolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cerebrolysin (Active Comparator): IV
  Interventions: Drug: cerebrolysin
- L-Alpha glycerylphosphorylcholine (Active Comparator): IV
  Interventions: Drug: L-Alpha glycerylphosphorylcholine
- citicoline (Active Comparator): IV and per os
  Interventions: Drug: citicoline

INTERVENTIONS:
Drug: citicoline — citicoline IV 2000 mg, then citicoline 900 mg/day (300mg*3 times per day) per os
  Arms: citicoline
Drug: L-Alpha glycerylphosphorylcholine — choline alfoscerate IV 1000mg daily 10 days
  Arms: L-Alpha glycerylphosphorylcholine
Drug: cerebrolysin — Cerebrolysin IV 10 ml daily 10 days
  Arms: cerebrolysin

SUMMARY:
Ischemic stroke (IS) causes high mortality and severe disability. To improve outcome it's very important to choose the right way of the management of the patient and an appropriate drugs.

There is a large number of the so-called neuroprotective drugs, which were effective in laboratory, but didn't show positive results in clinical studies with using traditional clinical scales scores as a primary outcome measures.

Specialists suggest, that the investigators could receive better results if the investigators change design of the studies, particularly if the investigators select more precise and sensitive method of assessment.

Aim of this study: to determine the role of navigated brain stimulation (NBS) for evaluation of the changes in the motor centers and motor tracts after administration of different cerebroprotective drugs. (The substances won't be compared to each other).

ELIGIBILITY:
Inclusion Criteria:

* patients from 3 to 6 months after ischemic stroke
* hemispheric infarction
* paresis from 2 to 4 scores by Medical Research Council Weakness Scale (MRC)

Exclusion Criteria:

* history of seizures
* pregnancy, lactation
* cognitive deficiency (poor compliance)
* acute renal failure
* acute hepatic failure
* oncological history
* cardiac pacemakers and other metal implants
* regular intake of any nootropic drugs
* Modified Ashford Scale scores 3 and more
* regular intake of anticonvulsants, neuromuscular relaxants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
MEP(motor evoked potential) parameter: motor threshold | 2 months
MEP(motor evoked potential) parameter: latency | 2 months
MEP(motor evoked potential) parameter: amplitude | 2 months

SECONDARY OUTCOMES:
Medical Research Council (MRC) Scale for Muscle Strength scores | 2 months
Barthel index | 2 months
Modified Rankin Scale (mRS) | 2 months
Number of Participants with Adverse Events | 2 months
Change from Baseline in Alpha waves percentage | 2 months
  EEG parameter
Change from Baseline in Beta waves percentage | 2 months
  EEG parameters
Change from Baseline in Delta waves percentage | 2 months
  EEG parameter
Change from Baseline in Theta waves percentage | 2 months
  EEG parameter
Presence of the abnormal epileptiform activity | 2 months
  EEG parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Institute of Brain, Yekaterinburg, Sverdlovsk Oblast, Russia